CLINICAL TRIAL: NCT03274986
Title: A Prospective, Randomized, Controlled, Multi-Center Clinical Study of the ACRYSOF® IQ Extended Depth of Focus IOL
Brief Title: A Clinical Study of the ACRYSOF® IQ Extended Depth of Focus Intraocular Lens (IOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILI875-C002
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- DFT015 (Experimental): ACRYSOF® IQ Extended Depth of Focus Intraocular lens (IOL), bilateral implantation
  Interventions: Device: ACRYSOF® IQ Extended Depth of Focus IOL; Procedure: Cataract surgery
- SN60WF (Active Comparator): ACRYSOF® IQ Monofocal IOL, bilateral implantation
  Interventions: Device: ACRYSOF® IQ Monofocal IOL; Procedure: Cataract surgery

INTERVENTIONS:
Device: ACRYSOF® IQ Extended Depth of Focus IOL — Implantable IOL intending to extend the depth of focus and provide continuous functional vision from distance to near while maintaining distance vision and a visual disturbance profile comparable to a monofocal IOL.
  Other Names: Model DFT015
  Arms: DFT015
Device: ACRYSOF® IQ Monofocal IOL — Monofocal IOL implanted for long-term use over the lifetime of the pseudophakic subject
  Other Names: Model SN60WF
  Arms: SN60WF
Procedure: Cataract surgery — IOL bilateral implantation

SUMMARY:
The purpose of the study is to demonstrate the safety and performance of ACRYSOF IQ extended depth of focus (EDF) intraocular lens (IOL) at Month 6. Depth of focus (DOF) is the amount of focal plane displacement behind a lens that does not degrade the image quality of a distant object. A larger DOF allows sharp images of closer objects and may provide improved vision at intermediate and near distances.

DETAILED DESCRIPTION:
Both eyes of a subject must require cataract surgery to qualify for enrollment into this study. Subjects participating in the trial will attend a total of 9 scheduled study visits over a 7-8 month period. Of the 9 visits, 1 is preoperative, 2 are operative, and the remaining 6 are postoperative visits. Primary endpoint data will be collected at the Month 6 (Day 120-180) post second eye implantation visit.

ELIGIBILITY:
Inclusion Criteria:

* Best Corrected Distance Visual Acuity (BCDVA) of 0.3 logarithm of the minimum angle of resolution (logMAR) (20/40 Snellen) or worse either with or without a glare source present (e.g., Brightness Acuity Tester)
* Preoperative regular astigmatism of < 1.0 D in both eyes
* Clear intraocular media other than cataract
* Diagnosed with cataract in both eyes
* Planned cataract removal by routine small incision surgery
* Calculated lens power between 18.0 and 25.0 diopter (D) [when targeted for emmetropia (0.0 D)]
* Willing and able to complete all required postoperative visits
* Able to comprehend and sign an ethics committee-approved statement of informed consent
* Potential postoperative BCDVA of 0.2 logMAR (20/32 Snellen) or better in each eye based on Investigator's medical opinion.

Exclusion Criteria:

* History of eye pathology and/or inflammation, as specified in the protocol
* Clinically significant/severe ocular surface disease that would affect study measurements based on Investigator expert medical opinion
* History of previous intraocular or corneal surgery
* Pregnant/lactating or has another condition with associated fluctuation of hormones that could lead to refractive changes
* Taking systemic medications that in the Investigator's best medical judgment may confound the outcome or increase the risk to the subject.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Research, Study Director — Alcon Research
Locations (11):
- United States (11):
  - Alcon Investigative Site, Birmingham, Alabama
  - Alcon Investigative Site, Fort Collins, Colorado
  - Alcon Investigative Site, Bradenton, Florida
  - Alcon Investigative Site, Sebring, Florida
  - Alcon Investigative Site, Gainesville, Georgia
  - Alcon Investigative Site, Rock Island, Illinois
  - Alcon Investigative Site, Cincinnati, Ohio
  - Alcon Investigative Site, Allenwood, Pennsylvania
  - Alcon Investigative Site, Kingston, Pennsylvania
  - Alcon Investigative Site, West Mifflin, Pennsylvania
  - Alcon Investigative Site, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCabe C, Berdahl J, Reiser H, Newsom TH, Cibik L, Koch D, Lemp-Hull J, Jasti S. Clinical outcomes in a U.S. registration study of a new EDOF intraocular lens with a nondiffractive design. J Cataract Refract Surg. 2022 Nov 1;48(11):1297-1304. doi: 10.1097/j.jcrs.0000000000000978. Epub 2022 May 26. PMID 35616507

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 11 investigative sites located in the United States.
Pre-assignment Details: 21 subjects discontinued prior to randomization, and 1 subject discontinued after randomization but prior to attempted implantation. This reporting group includes all subjects with attempted implantation, as treated. Note: 1 subject randomized to DFT015 was implanted with SN60WF. Subject withdrew at the 1 month visit.
Groups:
- DFT015: ACRYSOF® IQ Extended Depth of Focus IOL, bilateral implantation
Period: Overall Study
Arm/Group | DFT015 | SN60WF
Started (All subjects with attempted implantation, as treated.) | 107 | 113
Successful Implantation, as Treated | 107 | 113
Completed | 107 | 111
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population included all randomized eyes with successful IOL implantation (All-Implanted Analysis Set), as treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | DFT015 | SN60WF | Total
Number analyzed (Participants) | 107 | 113 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (7.82) | 68.8 (6.63) | 68.8 (7.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 64 | 123
  Male | 48 | 49 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 104 | 111 | 215
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 105 | 110 | 215
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Monocular Photopic Distance Corrected Intermediate Visual Acuity (DCIVA) [(Logarithm of the Minimum Angle of Resolution (logMAR)] 66 Centimeters (cm) From Spectacle Plane
Description: Visual acuity (VA) was tested monocularly (each eye separately) under photopic (well-lit) conditions using best distance correction adjusted for optical infinity, electronic Early Treatment Diabetic Retinopathy Study (ETDRS) charts at a distance of 66 cm from the spectacle plane. DCIVA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter or 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represented better VA. This analysis was prespecified for the first operative eye.
Time Frame: Month 6 (120-180 days post second eye implantation)
Population: All-Implanted Analysis Set, as treated
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 107 | 111
Number analyzed (Eyes) | 107 | 111
logMAR | 0.148 (0.0120) | 0.312 (0.0118)
Statistical Analysis 1: Comparison: DFT015 vs SN60WF; Test type: Superiority; p < 0.001, t-test, 2 sided — 2-sided p-value reported. A hypothesis test was based on a two sample t-test, with a type I error rate of 0.025, 1-sided; Least Squares Mean Difference = -0.164, 95% CI 2-sided [-0.197 to -0.131], Standard Error of Mean 0.0168 — Least squares mean difference (DFT015 - SN60WF)

2. Primary Outcome: Monocular Photopic Best Corrected Distance Visual Acuity (BCDVA) logMAR [(4 Meters (m)] From Spectacle Plane
Description: VA was tested monocularly under photopic conditions using the correction obtained from the best correction and no optical infinity adjustment, electronic ETDRS charts at a distance of 4 m from the spectacle plane. VA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter or 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represented better VA. This analysis was prespecified for the first operative eye.
Time Frame: Month 6 (120-180 days post second eye implantation)
Population: All-Implanted Analysis Set, as treated
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 107 | 111
Number analyzed (Eyes) | 107 | 111
logMAR | 0.016 (0.0091) | -0.036 (0.0089)
Statistical Analysis 1: Comparison: DFT015 vs SN60WF; Test type: Non-Inferiority — Non-Inferiority margin was 0.1 logMAR; t-test, 2 sided — The hypothesis test was based on a two-sample t-test, with a type I error rate of 0.05, 1-sided; Least Squares Mean Difference = 0.052, 95% CI 1-sided [upper limit 0.073], Standard Error of Mean 0.0127 — Least squares mean difference (DFT015 - SN60WF). The 1-sided 95% Upper Confidence Limit is presented

3. Primary Outcome: Monocular Depth of Focus (Measured in the Negative Direction From 0) at 0.20 logMAR From the Mean Defocus Curve
Description: Depth of focus was assessed at 4 meters under photopic (well-lit) conditions using best corrected distance refraction and added defocus. The depth of focus was estimated as the dioptric range between zero defocus and the first point on the negative lens induced mean defocus curve that crosses the 0.2 logMAR using a linear interpolation. A lower numeric value represents better VA. This analysis was pre-specified for the first operative eye. No formal statistical hypothesis testing was planned.
Time Frame: Month 6 (120-180 days post second eye implantation)
Population: All-Implanted Analysis Set, as treated. Number analyzed is the number of subjects/eyes with data available for analysis at specified defocus.
Measure: Number; unit: diopter
Units Other Than Participants: Eyes
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 107 | 111
Number analyzed (Eyes) | 107 | 111
diopter | 1.53 | 0.99
Statistical Analysis 1: Comparison: DFT015 vs SN60WF; Test type: Other; Hypothesis testing was not pre-specified; Difference in depth of focus = 0.54 — Difference in depth of focus (DFT015 - SN60WF)

4. Primary Outcome: Percentage of Eyes Achieving Monocular Photopic DCIVA 0.20 logMAR or Better
Description: VA was tested monocularly under photopic conditions using best distance correction adjusted for optical infinity, electronic ETDRS charts at a distance of 66 cm from the eye. DCIVA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter or 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represented better VA. This analysis was prespecified for the first operative eye. No formal statistical hypothesis testing was planned.
Time Frame: Month 6 (120-180 days post second eye implantation)
Population: All-Implanted Analysis Set, as treated.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 107 | 111
Number analyzed (Eyes) | 107 | 111
percentage of eyes | 72.9 | 25.2

5. Primary Outcome: Percentage of Subjects With Ocular Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device (test article). Ocular AEs are events localized to the eye. Cumulative and persistent serious adverse events as defined in ISO 11979-7:2014 were collected. This outcome measure was prespecified for the Model DFT015 first and second eyes. No formal statistical hypothesis testing was planned.
Time Frame: Day 0 (first operative eye visit), up to Month 6 (120-180 days post second eye implantation)
Population: This analysis population included all eyes with attempted IOL implantation (successful or aborted after contact with the eye) (Safety Analysis Set).
Measure: Number; unit: percentage of subjects
Units Other Than Participants: Eyes
Groups:
- DFT015 First Eye: All eyes with attempted test article implantation (successful or aborted after contact with the eye) in the first implanted eye
- DFT015 Second Eye: All eyes with attempted test article implantation (successful or aborted after contact with the eye) in the second implanted eye
Arm/Group | DFT015 First Eye | DFT015 Second Eye
Number analyzed (Participants) | 107 | 106
Number analyzed (Eyes) | 107 | 106
percentage of subjects
  Cumulative: Cystoid macular oedema | 0.9 | 0.0
  Cumulative: Hypopyon | 0.0 | 0.0
  Cumulative: Endophthalmitis | 0.0 | 0.0
  Cumulative: Lens dislocated from posterior chamber | 0.0 | 0.0
  Cumulative: Pupillary block | 0.0 | 0.0
  Cumulative: Retinal detachment | 0.0 | 0.0
  Cumulative: Secondary surgical intervention | 0.0 | 1.9
  Cumulative: Cataract operation complication | 0.0 | 1.9
  Cumulative: Hyphaema | 0.9 | 0.0
  Cumulative: Transient ischaemic attack | 0.9 | 0.0
  Persistent: Corneal stroma oedema | 0.0 | 0.0
  Persistent: Cystoid macular oedema | 0.0 | 0.0
  Persistent: Iritis | 0.0 | 0.0
  Persistent: Raised IOP requiring treatment | 0.0 | 0.0

6. Primary Outcome: Mesopic Contrast Sensitivity
Description: Contrast sensitivity (i.e., the ability to detect objects by distinguishing them from their background) was assessed monocularly with the subject's best spectacle correction under mesopic (low, but not quite dark) conditions at a distance of 8 (2.45 m) feet from the eye at a spatial frequency of 1.5, 3, 6, and 12 cycles per degree (cpd) using the Vector Vision CSV 1000-HGT with and without a glare source. Raw scores from contrast sensitivity testing were transformed to log units. A higher numeric value represented better contrast sensitivity. This analysis was prespecified for the first operative eye. No formal statistical hypothesis testing was planned.
Time Frame: Month 6 (120-180 days post second eye implantation)
Population: Safety Analysis Set. Number analyzed is the number of subjects/eyes with data available for analysis at without glare and with glare assessments.
Measure: Mean (Standard Deviation); unit: log unit
Units Other Than Participants: Eyes
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 107 | 113
Number analyzed (Eyes) | 107 | 113
log unit
  1.5 cpd Without Glare: number analyzed (Participants) | 107 | 111
  1.5 cpd Without Glare: number analyzed (Eyes) | 107 | 111
  1.5 cpd Without Glare | 1.506 (0.2560) | 1.498 (0.2434)
  3 cpd Without Glare: number analyzed (Participants) | 107 | 111
  3 cpd Without Glare: number analyzed (Eyes) | 107 | 111
  3 cpd Without Glare | 1.447 (0.3381) | 1.482 (0.2829)
  6 cpd Without Glare: number analyzed (Participants) | 107 | 111
  6 cpd Without Glare: number analyzed (Eyes) | 107 | 111
  6 cpd Without Glare | 1.340 (0.3850) | 1.548 (0.3177)
  12 cpd Without Glare: number analyzed (Participants) | 107 | 111
  12 cpd Without Glare: number analyzed (Eyes) | 107 | 111
  12 cpd Without Glare | 0.840 (0.3681) | 1.003 (0.3769)
  1.5 cpd With Glare: number analyzed (Participants) | 107 | 111
  1.5 cpd With Glare: number analyzed (Eyes) | 107 | 111
  1.5 cpd With Glare | 1.504 (0.2555) | 1.475 (0.2569)
  3 cpd With Glare: number analyzed (Participants) | 107 | 111
  3 cpd With Glare: number analyzed (Eyes) | 107 | 111
  3 cpd With Glare | 1.458 (0.3304) | 1.499 (0.2838)
  6 cpd With Glare: number analyzed (Participants) | 107 | 111
  6 cpd With Glare: number analyzed (Eyes) | 107 | 111
  6 cpd With Glare | 1.364 (0.3856) | 1.529 (0.3256)
  12 cpd With Glare: number analyzed (Participants) | 107 | 111
  12 cpd With Glare: number analyzed (Eyes) | 107 | 111
  12 cpd With Glare | 0.817 (0.3494) | 0.999 (0.4020)

7. Secondary Outcome: Monocular Photopic Distance Corrected Near Visual Acuity (DCNVA) (logMAR) 40 cm From Spectacle Plane
Description: VA was tested monocularly under photopic conditions using best distance correction adjusted for optical infinity, electronic ETDRS chart set at 40 cm from the spectacle plane. VA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter or 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represented better VA. This analysis was prespecified for the first operative eye.
Time Frame: Month 6 (120-180 days post second eye implantation)
Population: All-Implanted Analysis Set, as treated.
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 107 | 111
Number analyzed (Eyes) | 107 | 111
logMAR | 0.359 (0.0147) | 0.515 (0.0144)
Statistical Analysis 1: Comparison: DFT015 vs SN60WF; Test type: Superiority; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.156, 95% CI 2-sided [-0.197 to -0.115], Standard Error of Mean 0.0206 — Least squares mean difference (DFT015 - SN60WF)

8. Secondary Outcome: Percentage of Subjects Who Respond "Never" to Question 1 of the Intraocular Lens Satisfaction (IOLSAT) Questionnaire: "Overall, in the Past 7 Days, How Often Did You Need to Wear Eyeglasses to See?"
Description: The IOLSAT questionnaire assessed the subjective quality of vision with respect to need for spectacles, as well as the subject's expectation and satisfaction with their quality of vision at 6 months. Results are reported consistent with multiple testing strategy.
Time Frame: Month 6 (120-180 days post second eye implantation)
Population: All-Implanted Analysis Set, as treated.
Measure: Number; unit: percentage of subjects
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 102 | 111
percentage of subjects | 21.6 | 3.6
Statistical Analysis 1: Comparison: DFT015 vs SN60WF; Test type: Other; Difference in percentage = 18, 95% CI 2-sided [9.65 to 27.37] — 95% CI for the difference (DFT015 - SN60WF) is estimated using Miettinen-Nurminen method (1985)

9. Secondary Outcome: Monocular Photopic Uncorrected Intermediate Visual Acuity (UCIVA) (logMAR) 66 cm From Spectacle Plane
Description: VA was tested monocularly under photopic conditions with no refractive correction or adjustment for optical infinity, using electronic ETDRS charts at a distance of 66 cm from the spectacle plane. UCIVA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter or 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represented better VA. This analysis was prespecified for the first operative eye. No formal statistical hypothesis testing was planned.
Time Frame: Month 6 (120-180 days post second eye implantation)
Population: All-Implanted Analysis Set, as treated.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 107 | 111
Number analyzed (Eyes) | 107 | 111
logMAR | 0.136 (0.110) | 0.261 (0.147)

10. Secondary Outcome: Monocular Photopic Uncorrected Distance Visual Acuity (UCDVA) (logMAR)
Description: VA was tested monocularly under photopic conditions without refractive correction but with adjustment for optical infinity, electronic ETDRS charts at a distance of 4 m from the eye. +0.25 D spherical power was applied to correct for optical infinity. UCDVA was measured in logMAR, with 0.02 logMAR increment corresponding to a single letter or 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represented better VA.This analysis was prespecified for the first operative eye. No formal statistical hypothesis testing was planned.
Time Frame: Month 6 (120-180 days post second eye implantation)
Population: All-Implanted Analysis Set, as treated.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 107 | 111
Number analyzed (Eyes) | 107 | 111
logMAR | 0.117 (0.122) | 0.056 (0.148)

11. Secondary Outcome: Percentage of Subjects With Visual Disturbances as Reported by the Subjects Using the Questionnaire for Visual Disturbances (QUVID)
Description: Rates of severe and most bothersome visual disturbances as reported by the subjects on the QUVID questionnaire, a Patient Reported Outcome (PRO) questionnaire. No formal statistical hypothesis testing was planned.
Time Frame: Month 6 (120-180 days post second eye implantation)
Population: Safety Analysis Set. Number analyzed is the number of subjects/eyes with data available for analysis at specified visual disturbances.
Measure: Number; unit: percentage of subjects
Arm/Group | DFT015 | SN60WF
Number analyzed (Participants) | 106 | 113
percentage of subjects
  Severe: Starbursts: number analyzed (Participants) | 106 | 110
  Severe: Starbursts | 3.8 | 2.7
  Severe: Halos: number analyzed (Participants) | 106 | 110
  Severe: Halos | 0.9 | 0.9
  Severe: Glare: number analyzed (Participants) | 105 | 111
  Severe: Glare | 0.0 | 0.0
  Severe: Hazy vision: number analyzed (Participants) | 105 | 111
  Severe: Hazy vision | 0.0 | 0.0
  Severe: Blurred vision: number analyzed (Participants) | 106 | 111
  Severe: Blurred vision | 0.0 | 0.0
  Severe: Double vision: number analyzed (Participants) | 106 | 111
  Severe: Double vision | 0.0 | 0.0
  Severe: Dark area: number analyzed (Participants) | 106 | 111
  Severe: Dark area | 0.9 | 0.9
  Most Bothersome: Starbursts: number analyzed (Participants) | 106 | 110
  Most Bothersome: Starbursts | 1.9 | 0.9
  Most Bothersome: Halos: number analyzed (Participants) | 106 | 110
  Most Bothersome: Halos | 0.9 | 0.0
  Most Bothersome: Glare: number analyzed (Participants) | 105 | 111
  Most Bothersome: Glare | 0.0 | 0.0
  Most Bothersome: Hazy vision: number analyzed (Participants) | 105 | 111
  Most Bothersome: Hazy vision | 0.0 | 0.0
  Most Bothersome: Blurred vision: number analyzed (Participants) | 106 | 111
  Most Bothersome: Blurred vision | 0.9 | 1.8
  Most Bothersome: Double vision: number analyzed (Participants) | 106 | 111
  Most Bothersome: Double vision | 0.0 | 0.0
  Most Bothersome: Dark area: number analyzed (Participants) | 106 | 111
  Most Bothersome: Dark area | 0.9 | 0.9

ADVERSE EVENTS:
Time Frame: Pre-operation (Day -28) up to Day 120-180 (post second eye implantation), up to 8 months
Description: An AE was any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the investigational medical device. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. Safety Analysis Set. "At Risk" population of preoperative and systemic AEs is reported in units of subjects; all other AE populations are reported in units of eyes.
Groups:
- Preoperative: All subjects in the safety analysis set prior to initiation of treatment
- DFT015 Systemic: All subjects with attempted test article implantation (successful or aborted after contact with the eye)
- SN60WF First Eye: All eyes with attempted control article implantation (successful or aborted after contact with the eye) in the first implanted eye
- SN60WF Second Eye: All eyes with attempted control article implantation (successful or aborted after contact with the eye) in the second implanted eye
- SN60WF Systemic: All subjects with attempted control article implantation (successful or aborted after contact with the eye)
Arm/Group | Preoperative | DFT015 First Eye | DFT015 Second Eye | DFT015 Systemic | SN60WF First Eye | SN60WF Second Eye | SN60WF Systemic
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/107 | 0/106 | 0/107 | 0/113 | 0/113 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/220 | 3/107 | 2/106 | 7/107 | 3/113 | 1/113 | 4/113
Other Adverse Events (participants affected / at risk) | 0/220 | 5/107 | 6/106 | 0/107 | 9/113 | 8/113 | 0/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preoperative (N=220) | DFT015 First Eye (N=107) | DFT015 Second Eye (N=106) | DFT015 Systemic (N=107) | SN60WF First Eye (N=113) | SN60WF Second Eye (N=113) | SN60WF Systemic (N=113)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Heart valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystoid macular oedema (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ulcer haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Bladder injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Surgical procedure repeated (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aneurysm repair (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lens extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitrectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyphaema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Preoperative (N=220) | DFT015 First Eye (N=107) | DFT015 Second Eye (N=106) | DFT015 Systemic (N=107) | SN60WF First Eye (N=113) | SN60WF Second Eye (N=113) | SN60WF Systemic (N=113)
Posterior capsule opacification (Eye disorders) | 0 | 5 | 6 | 0 | 9 | 8 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT03274986/SAP_000.pdf
  • Study Protocol (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT03274986/Prot_001.pdf